CLINICAL TRIAL: NCT07004868
Title: Inflammation, Cachexia and Therapeutic Response in Lung Cancer Treated With Immune Checkpoint Inhibitors: Exploratory Observational Study
Acronym: LCab
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR240341 - LCab
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer (NSCLC)
Keywords: immune checkpoint inhibitors; inflammation; cachexia
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Inflammation; Cachexia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is the leading cause of cancer-related death in France and globally, with 2.48 million new cases diagnosed in 2022, accounting for nearly 13% of global cancer incidence. Despite recent advances, it remains a major health issue due to late-stage diagnosis and high patient and societal burden. New insights into tumor and immune pathways have led to the development of targeted therapies, including tyrosine kinase inhibitors and therapeutic antibodies. Among these, immune checkpoint inhibitors (ICIs) such as nivolumab, pembrolizumab, atezolizumab, and durvalumab have significantly improved outcomes for some patients by reactivating T-cell responses.

The LCAb (Lung Cancer Antibodies) research project focuses on studying the interindividual variability of clinical response to ICI in lung cancer. These therapies are now used across various lung cancer types and stages, including early and advanced disease. Most ICIs are administered at fixed doses, without considering patient-specific factors as blood concentrations, tumor burden, body weight or nutritional status. The study hypothesizes that fixed dosing may affect treatment response and survival outcomes, highlighting the need for more personalized approaches.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death in France and worldwide. Its incidence is significant, with 2.48 million new cases diagnosed in 2022, representing nearly 13% of the total global cancer incidence. Despite recent therapeutic advances, it remains a major public health issue due to its frequent diagnosis at a metastatic stage, which results in high morbidity and mortality for patients and significant costs for society.

A better understanding of tumor and immune signaling pathways has recently led to the discovery of new molecular targets, such as immune checkpoints. The therapeutic arsenal against lung cancer has thus expanded to include new molecules such as tyrosine kinase inhibitors and therapeutic antibodies (Abs). The latter represent the majority of anticancer biotherapies, with more than 50 approved agents for solid or hematologic cancers.

In particular, antibodies targeting immune checkpoints (ICIs - immune checkpoint inhibitors), such as nivolumab, pembrolizumab, atezolizumab, and durvalumab, have revolutionized the management of certain lung cancer patients by reversing T-cell exhaustion, allowing some of them to become long-term responders.

The research project "Pharmacokinetics of Immune Checkpoint Inhibitor Antibodies Used in Lung Cancer" (LCAb - Lung Cancer Antibodies) aims to study the blood concentrations and pharmacokinetics of various ICI-type antibodies used in the treatment of lung cancer.

Lung cancer is characterized by multiple histological types, stages, and molecular profiles, each associated with different therapeutic options. ICI-type antibodies have numerous indications in lung cancer, and these indications have continued to expand in recent years. They are now used not only in metastatic stages but also in localized and locally advanced stages. These molecules have led to a marked improvement in the prognosis of lung cancer patients. However, their effectiveness varies from one patient to another.

The study focuses on anti-PD-1 and anti-PD-L1 ICI antibodies used routinely in lung cancer, regardless of histology or stage, whether administered alone or in combination with chemotherapy. Most of these antibodies are administered at a fixed dose, without adjustment for age, weight, general health, or nutritional status of the patients.We hypothesize that the use of fixed-dose ICIs in lung cancer may influence therapeutic response and patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Diagnosis of lung cancer, any histology, any stage
* Treatment with Ab ICI, with or without chemotherapy
* 1st administration of Ab ICI

Exclusion Criteria:

* Patient not followed at the CHRU de Tours
* Person under protective supervision
* Opposition to data processing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a lung cancer treated with immune checkpoint inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
time to progression | Month 36
  time between 1st administration of Ab ICI and progression or death from any cause.

SECONDARY OUTCOMES:
weight | from day 0 to month 36 at each patient visit
Serum CRP concentration | from day 0 to month 36 at each patient visit
Serum Ab ICI concentration | from day 0 to month 36 at each patient visit
  measured using validated ELISA (Enzyme-Linked Immunosorbent Assay) techniques
Drug toxicity | from day 0 to month 36 at each patient visit
Overall survival | from day 0 to month 36 at each patient visit
  time between first administration of Ab ICI and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Marion FERREIRA, Dr, Principal Investigator — University Hospital, Tours
Locations (1):
- university hospital, Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided